CLINICAL TRIAL: NCT02932137
Title: Potential Effect of Anti-infection by Low-dose IL-2 in Treatment of SLE
Brief Title: Anti-infection of Low-does IL-2 in SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Professor and chief of department of rheumatology and immunology, Peking University People's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IL-2-20160505
Record Dates: First submitted 2016-10-08; First posted 2016-10-13 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE,IL-2
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interleukin-2 (Experimental): Interleukin-2 to treat activated SLE.
  Interventions: Drug: Interleukin-2
- Traditional therapy (No Intervention): Treat activated SLE with glucocorticoid or immunosuppressor.

INTERVENTIONS:
Drug: Interleukin-2 — Patients receive low dose recombinant human Interleukin-2（HrIL-2）
  Other Names: Recombinant Human Interleukin-2,125Ala, SL Pharm
  Arms: Interleukin-2

SUMMARY:
The objective of this clinical study is to evaluate the potential effect of anti-infection of low-does IL-2 in patients with SLE.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune syndrome affecting various organs.Many feel that glucocorticoid and immunosuppressor are the standard therapy for patients with SLE. While it can improve the risk of infection among SLE patients. A novel therapy to treat SLE with low-does IL-2 has been identified recently. IL-2 also used to against some virus infect. So we hypothesized that low-dose IL-2 could reduce risk of infection in SLE patients.

Methods: A total of SLE patients (n=30) were divided into two groups randomly. One received standard therapy, while another one administrate with low-does IL-2 plus standard therapy.Each patient will be treated with low-dose IL-2. The end points are clinical and immunologic response.

Expected Results: This trail wlii provide both clinical and basic profe that low-dose IL-2 plus standard therapy have lower infection risk in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology criteria for the diagnosis of SLE.
* Under standard treatment (≥ 2 months) at the time of inclusion
* Background treatment failed to control flares or to permit prednisone tapering
* With at least one of the following manifestations: thrombocytopenia, disease-associated rash, mouth ulcer, non-infectious type of fever, active vasculitis, renal disorder(proteinuria>0.5g/day), neuropsychiatric SLE.
* Positive for at least one of the following laboratory tests: ANA>1:160, anti-dsDNA, immunoglobulin>20g/L, decreased C3 or C4, leukopenia<3×10^9/L, thrombocytopenia<100×10^9/L;
* SLE disease activity index(SLEDAI) ≥ 8.
* Negative HIV test.
* Negative for hepatitis B and C virus.
* Written informed consent form.

Exclusion Criteria:

* Sever chronic liver, kidney, lung or heart dysfunction; (heart failure (≥ grade III NYHA), hepatic insufficiency (transaminases> 3N) )
* Serious infection such as bacteremia, sepsis;
* Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or Basocellular carcinoma);
* High-dose steroid pulse therapy (>1.5mg/kg) or IV bolus of corticosteroids in the last 2 months.
* History of administration of rituximab or other biologics;
* Purified protein derivative (tuberculin) >10mm
* Mental disorder or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give information;
* Inability to comply with IL-2 treatment regimen.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Immunological Responses | week 0 and week 10
  The increased intracellular factors which could reflect the organic immunity

SECONDARY OUTCOMES:
Virus titers | week 0 and week 10
  The reduced titers of virus in SLE patients

OTHER OUTCOMES:
SLEDAI Score | week 0 and week 10
  Assessment version of the SLE Disease Activity Index (SELENA-SLEDAI) change.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD and PhD, Principal Investigator — Peking University Institute of Rheumatology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] He J, Zhang R, Shao M, Zhao X, Miao M, Chen J, Liu J, Zhang X, Zhang X, Jin Y, Wang Y, Zhang S, Zhu L, Jacob A, Jia R, You X, Li X, Li C, Zhou Y, Yang Y, Ye H, Liu Y, Su Y, Shen N, Alexander J, Guo J, Ambrus J, Lin X, Yu D, Sun X, Li Z. Efficacy and safety of low-dose IL-2 in the treatment of systemic lupus erythematosus: a randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2020 Jan;79(1):141-149. doi: 10.1136/annrheumdis-2019-215396. Epub 2019 Sep 19. PMID 31537547